CLINICAL TRIAL: NCT04622683
Title: Effects of Hepatic Ultrasound on Metabolic Homeostasis
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2000026135
Record Dates: First submitted 2020-11-02; First posted 2020-11-10 (Actual); Last update posted 2024-12-16 (Actual); Status verified 2024-12

CONDITIONS: Healthy; Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — High-Energy Shock Waves

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Control Group- Healthy, Lean Individuals (Experimental): Determine whether ultrasound exposure at the porta hepatis will affect plasma glucose levels in lean, healthy control subjects.
  Interventions: Procedure: Ultrasound
- Overweight/obese individuals who have normal glucose tolerance or impaired glucose tolerance (Active Comparator): Determine whether three episodes of porta hepatic ultrasound exposure will affect plasma glucose levels as well as insulin sensitivity among overweight/obese individuals who have normal glucose tolerance or impaired glucose tolerance (as defined by OGTT.
  Interventions: Procedure: Ultrasound

INTERVENTIONS:
Procedure: Ultrasound — To determine whether ultrasound exposure at the porta hepatis will affect plasma glucose levels. To also determine whether porta hepatic ultrasound exposure will affect plasma glucose levels as well as insulin sensitivity among overweight/obese individuals who have normal glucose tolerance or impaired glucose tolerance (as defined by OGTT.

SUMMARY:
The purpose of this study is to define the effect of ultrasound exposure of the liver in the region of the porta hepatis on glucose homeostasis and insulin resistance in healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

* 18 - 60 years of age
* Aim 1: Healthy lean men and women, BMI<24 kg/m2, with normal fasting glucose (blood glucose between 60 and 100mg/dl and normal glucose tolerance on OGTT (blood glucose <140 mg/dl at 2 hours post glucose challenge) at the screening visit.
* Aim 2: Overweight and obese men and women, BMI 25 - 35 kg/m2

Exclusion Criteria:

* Type 1 and type 2 diabetes
* Surgery in the past 90 days
* Previous surgery of the spleen or splenectomy, esophagus, lungs, stomach, duodenum, or liver
* Recent traumatic injury, including intra-cerebral hemorrhage and visceral injury
* End stage renal disease and/or uremia
* Active malignancy
* Previous leukemia and/or lymphoma
* Human immunodeficiency virus infection or AIDS
* Rheumatoid arthritis or other immune-mediated diseases (e.g. inflammatory bowel disease)
* Arrhythmias, including but not limited to, atrial fibrillation, atrial flutter, bradycardia, ventricular arrhythmias, and A-V block
* Implanted pacemaker or cardioverter/defibrillator (AICD)
* History of stable or unstable angina, myocardial infarction, angioplasty or coronary arterial by-pass grafting surgery
* History of stroke or TIA
* History of deep venous thrombosis (DVT) and/or pulmonary embolism (PE)
* Previous episodes of pancreatitis
* Spinal disorders
* Chronic pain syndromes
* History of thrombosis or bleeding disorders
* Stage III-IV pressure ulcers
* Sickle cell anemia or other anemia syndromes
* Monocytosis
* Thrombocytopenia
* Diagnosed with fever of unknown origin (FUO)
* Previously or currently implanted vagus nerve stimulator
* Previously or currently implanted spinal cord stimulator
* Other chronically-implanted electronic medical device
* History of seizures
* History of cancer
* Individuals who have taken any of the following medications within two weeks of receiving ultrasound delivery: anti-coagulant, anti-platelet, anti-inflammatory, immunosuppressive agents, alpha and/or beta adrenoceptor blocking agents, anti-seizure medications, anti-diabetic medication
* Individuals with a substance abuse problem
* Pregnant women
* Ascites detected in the abdomen that may effect delivery of shear wave elastroghapy pulse

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 37 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-09-13 (Actual); Study Completion 2023-09-13 (Actual)

PRIMARY OUTCOMES:
Insulin Resistance | 1 week
  Change in OGTT measurements after Hepatic Ultrasound

CONTACTS AND LOCATIONS:
Overall Officials: Raimund Herzog, MD, Principal Investigator — Yale University
Locations (1):
- Yale-New Haven Hospital, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
Upon request to Principal Investigator de-identified data can be requested.
Time Frame: Dependent upon request.
Access Criteria: Email to Principal Investigator

REFERENCES:
- [Background] Schwartz GJ. Roles for gut vagal sensory signals in determining energy availability and energy expenditure. Brain Res. 2018 Aug 15;1693(Pt B):151-153. doi: 10.1016/j.brainres.2018.04.004. PMID 29903617
- [Background] Cotero V, Fan Y, Tsaava T, Kressel AM, Hancu I, Fitzgerald P, Wallace K, Kaanumalle S, Graf J, Rigby W, Kao TJ, Roberts J, Bhushan C, Joel S, Coleman TR, Zanos S, Tracey KJ, Ashe J, Chavan SS, Puleo C. Noninvasive sub-organ ultrasound stimulation for targeted neuromodulation. Nat Commun. 2019 Mar 12;10(1):952. doi: 10.1038/s41467-019-08750-9. PMID 30862827